CLINICAL TRIAL: NCT01305252
Title: CombinatiON Up-FRON t Therapy for PAH - A Phase 4, Randomized, Multicenter Study of Inhaled Treprostinil in Treatment naïve Pulmonary Arterial Hypertension Patients Starting on Tadalafil
Brief Title: A 48-week Study of the Effect of Dual Therapy (Inhaled Treprostinil and Tadafafil) Versus Monotherapy (Tadalafil).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Roham T. Zamanian, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-07152010-6565; IRB protocol # 18305
Record Dates: First submitted 2010-11-02; First posted 2011-02-28 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tadalafil alone (Active Comparator): tadalafil 40mg QD(Tadalafil 20 mg QD PO increasing to 40 mg QD as tolerated).
  Interventions: Drug: tadalafil
- tadalafil and treprostinil inhalations (Active Comparator): Treprostinil inhalation QID starting at 3 breaths per inhalation & gradually increasing to 9 breaths.Each breath provides approximately 6 mcg of treprostinil.Tadalafil 20 mg QD PO increasing to 40 mg QD as tolerated.
  Interventions: Drug: treprostinil inhalations; Drug: tadalafil

INTERVENTIONS:
Drug: treprostinil inhalations — Treprostinil inhalation QID starting at 3 breaths per inhalation & gradually increasing to 9 breaths. Each breath provides approximately 6mcg of treprostinil.
  Other Names: Tyvaso
  Arms: tadalafil and treprostinil inhalations
Drug: tadalafil — tadalafil 20mg QD PO increasing to 40mg QD as tolerated
  Other Names: Adcirca

SUMMARY:
The Study Hypothesis:

Aggressive, upfront, dual therapy for treatment-naïve NYHA I/II/III PAH is superior to a traditional "step-up" approach.

The study will evaluate:

1. Impact of dual, upfront, therapy on cardiovascular parameters in PAH as gauged by cardiac magnetic resonance imaging (cMRI) at 24 weeks and event free survival at outcome at 48 weeks.
2. Value of novel biomarkers (NT-pro BNP, Mts1/S100A4, and insulin resistance) and cutting-edge imaging technologies (cardiac MRI) as newer endpoints for clinical trials in PAH.
3. Utility of longer clinical trial design with the use of combined clinical events as time to clinical worsening surrogate

DETAILED DESCRIPTION:
This is a 48 week interventional study evaluating the effect of Dual therapy ( Treprostinil inhalations and Tadalafil) versus Mono therapy (Tadalafil). The impact of the therapy on cardiovascular parameters in PAH measured at 24 weeks and event free survival outcome at 48 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 and < 75 years at baseline visit.
2. Diagnosis of Idiopathic PAH, Heritable PAH (including Hereditary Hemorrhagic Telangiectasia), Associated PAH (including collagen vascular disorders, drug+toxin exposure, repaired congenital heart disease repaired > 5 years, portopulmonary disease, and human immunodeficiency virus (HIV) infection not on protease inhibitor).
3. PAH treatment naïve including any prostacycline, endothelin receptor antagonist, or phosphodiesterase inhibitors within 12 months prior to enrollment.
4. Previous Right Heart Catheterization that documented:

   1. Mean PAP; 25 mmHg.
   2. Pulmonary capillary wedge pressure < 15 mmHg.
   3. Pulmonary Vascular Resistance; 3.0 Wood units or 240 dynes/sec/cm5 5.6MW distances; 150 m and < 450 meters.

6. WHO functional class II or III as judged by principal investigators.

Exclusion Criteria:

Exclusion criteria:

1. Group II - V pulmonary hypertension.
2. PAH with unrepaired congenital heart defect.
3. Current or prior PAH treatments within the last 6-12 months including experimental PAH therapies (including but not limited to tyrosine kinase inhibitors, rho-kinase inhibitors, phosphodiesterase inhibitors, prostacycline, or cGMP modulators).
4. TLC < 60% predicted; if TLC b/w 60 and 70% predicted, high resolution computed tomography must be available to exclude significant interstitial lung disease.
5. FEV1 / FVC < 70% predicted and FEV1 < 60% predicted
6. Significant left-sided heart disease (based on pre-trial Echocardiogram):

   1. Significant aortic or mitral valve disease
   2. Diastolic dysfunction ; Grade II C.LV systolic function < 45%

   d. Pericardial constriction e. Restrictive cardiomyopathy f. Significant coronary disease with demonstrable ischemia
7. Chronic renal insufficiency defined as an estimated creatinine clearance < 30 ml/min (by MDRD equation)
8. Current atrial arrhythmias
9. Uncontrolled systemic hypertension: SBP > 160 mm or DBP > 100mm
10. Severe hypotension: SBP < 80 mmHg.
11. Pregnant or breast-feeding
12. Psychiatric, addictive, or other disorder that compromises patient's ability to provide informed consent, follow study protocol, and adhere to treatment instructions
13. Co-morbid conditions that would impair a patient's exercise performance and ability to assess WHO functional class, including but not limited to chronic low-back pain or peripheral musculoskeletal problems.
14. Contraindications for magnetic resonance imaging, including significant claustrophobia, implanted metallic objects, or others as per Appendix X).
15. Known allergy to treprostinil or tadalafil.
16. Active oral nitrate use.
17. Diabetes mellitus.
18. Planned initiation of cardiac or pulmonary rehabilitation during period of study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roham T. Zamanian, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Northwestern University, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil Alone: tadalafil 40mg QD
  tadalafil: tadalafil 20mg QD PO increasing to 40mg QD as tolerated
- Tadalafil and Treprostinil Inhalations: inhaled treprostinil: Treprostinil inhalation QID starting at 3 breaths per inhalation & gradually increasing to 9 breaths. Each breath provides approximately 6mcg of treprostinil.
  tadalafil: tadalafil 20mg QD PO increasing to 40mg QD as tolerated
Period: Overall Study
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations
Started | 10 | 11
Completed | 9 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.4) | 52.1 (9.7) | 51.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricular Ejection Fraction
Description: Effect of dual-upfront therapies versus mono-therapy on percent change of right ventricular function assesed by cardiac MRI (cMRI) at 24 weeks compared with the baseline.
Time Frame: Basline and 24 weeks
Measure: Mean (Inter-Quartile Range); unit: percent change
Arm/Group | Tadalafil and Treprostinil Inhalations | Tadalafil Alone
Number analyzed (Participants) | 11 | 10
percent change | 7.45 [0.95 to 13.96] | 2.8 [-1.49 to 7.09]
Statistical Analysis 1: Comparison: Tadalafil and Treprostinil Inhalations; Test type: Superiority or Other; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Tadalafil Alone; Test type: Superiority or Other; p = 0.17, t-test, 2 sided

2. Secondary Outcome: 6 Minute Walk Distance
Description: Change in 6MWD during 24 week period compared between Tada and Tada+iTre.
Time Frame: Baseline and 24 weeks
Measure: Mean (Inter-Quartile Range); unit: meters
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations
Number analyzed (Participants) | 10 | 11
meters | 82.63 [23.40 to 141.86] | 87.69 [6.98 to 168.41]

3. Secondary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: Change from baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tadalafil and Treprostinil Inhalations | Tadalafil Alone
Number analyzed (Participants) | 11 | 10
pg/mL | 1239 (1393) | 988.4 (827.6)

4. Secondary Outcome: Change in NYHA/WHO Class
Description: At 48 week,WHO/NYHA functional class was assessed for change in WHO/NYHA functional class.Change NYHA is measured as decrease or increase in NYHA class in the subjects compared with baseline.
  NYHA /WHO functional class is described below:
  NYHA functional class I:no symptoms and no limitation in ordinary physical activity NYHA functional class II:Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity NYHA functional class III:Marked limitation in activity due to symptoms, even during less-than-ordinary activity NYHA functional class IV:Severe limitations. Experiences symptoms even while at rest A higher functional class represent worse symptoms.
Time Frame: Baseline and 48 week
Measure: Number; unit: participants
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations
Number analyzed (Participants) | 10 | 11
participants | 6 | 11
Statistical Analysis 1: Comparison: Tadalafil Alone; Test type: Superiority or Other; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Tadalafil and Treprostinil Inhalations; Test type: Superiority or Other; p = 0.33, t-test, 2 sided

5. Secondary Outcome: B-type Natriuretic Peptide (BNP)
Description: B-type Natriuretic peptide measures the percent change from baseline.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations
Number analyzed (Participants) | 10 | 11
percent change | 374 (133.8) | 295.6 (133.2)

ADVERSE EVENTS:
Time Frame: initial 24 weeks
Arm/Group | Tadalafil Alone | Tadalafil and Treprostinil Inhalations
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 9/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil Alone (N=10) | Tadalafil and Treprostinil Inhalations (N=11)
Death (Cardiac disorders) | 1 (1) | 0 (0) — Death attributed to septic shock and ensuring renal failure.Not clinically deemed to be related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil Alone (N=10) | Tadalafil and Treprostinil Inhalations (N=11)
Nasal congestion/allergic Rhinitis (General disorders) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 3
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Dental infection (Infections and infestations) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Edema (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations: small,2 center study,Placebo Un-blinded,Limited event rates/Time to clinical worsening and harmonization of measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No